CLINICAL TRIAL: NCT03084523
Title: Treatment Targets for Inflamed Intracranial Atherosclerosis on Vessel Wall MRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Adam de Havenon, Principle Investigator, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000031256
Record Dates: First submitted 2017-02-01; First posted 2017-03-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Intracranial Atherosclerosis
MeSH Terms: conditions — Stroke; Intracranial Arteriosclerosis | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 1 (Experimental): 80 patients with intracranial atherosclerosis
  Interventions: Drug: Ferumoxytol Injectable Product

INTERVENTIONS:
Drug: Ferumoxytol Injectable Product — Patients will be administered a single dose of ferumoxytol as an MRI contrast
  Other Names: Feraheme

SUMMARY:
Intracranial atherosclerosis (ICAS) accounts for 10 to 40%, depending on ethnicity, of the 700,000 ischemic strokes in the United States every year. The annual rate of recurrent stroke in patients with optimally treated ICAS remains more than twice the average of other stroke etiologies (12.5% vs. 5). A robust literature has established that vessel wall magnetic resonance imaging (vwMRI) of extracranial carotid vessel wall enhancement (VWE) can predict stroke, independent of stenosis. VWE has been reported in symptomatic ICAS, but the role of local and systemic inflammation is unknown. Inflammatory biomarkers are elevated in symptomatic extracranial atherosclerosis, but the association with vwMRI findings in ICAS has not yet been explored. VWE is typically demonstrated by the uptake of gadolinium MRI contrast into the aneurysm wall or atherosclerotic plaque. A novel MRI contrast agent, ferumoxytol, allows multi-contrast weighting on T1w and T2w images and provides important insight into the role of local vessel wall inflammation by accumulating in macrophages on delayed T2* sequences. To identify effective prevention and treatment strategies for cerebrovascular disease, we need to critically evaluate vwMRI techniques, determine VWE prevalence, and explore the link between VWE and inflammation.

DETAILED DESCRIPTION:
Intracranial atherosclerosis accounts for 10 to 40%, depending on ethnicity, of the 700,000 ischemic strokes in the United States every year.The annual rate of recurrent stroke in patients with optimally treated Intracranial atherosclerosis remains more than twice the average of other stroke etiologies (12.5% vs. 5%).A robust literature has established that vessel wall MRI of extracranial carotid vessel wall enhancement can predict stroke, independent of stenosis. Vessel wall enhancement has been reported in symptomatic intracranial atherosclerosis. Vessel wall enhancement is typically demonstrated by the uptake of gadolinium MRI contrast into the atherosclerotic plaque. A novel MRI contrast agent, ferumoxytol, allows multicontrast weighting on T1w and T2w images and provides important insight into the role of local vessel wall inflammation by accumulating in macrophages on delayed T2* sequences.

To identify effective prevention and treatment strategies for cerebrovascular disease, the investigator(s) need to critically evaluate vessel wall MRI techniques, determine vessel wall enhancement prevalence, and explore the link between vessel wall enhancement and inflammation. The investigator(s) hypothesize that vessel wall enhancement is reliable, associated with symptomatic Intracranial atherosclerosis. In order to answer our hypotheses, the investigator(s) propose a pilot study on 80 participants. The investigator(s) will opportunistically enroll participants who receive standard of care vessel wall MRI with gadolinium contrast or perform a baseline vessel wall MRI with gadolinium if needed. Intracranial atherosclerosis participants will have a total of 2-3 study vessel wall MRIs. Study MRI #1 will be performed with gadolinium, if a standard of care MRI has not already been performed. Study MRI #2 will be performed 72-78 hours post- using ferumoxytol contrast infusion. Study MRI #3 is a follow-up vessel wall MRI with gadolinium in 1 year.

ELIGIBILITY:
80 patients will be enrolled in this prospective cross-sectional study of Intracranial atherosclerosis.

* Inclusion Criteria:

  * intracranial atherosclerosis (stenosis ≥50%)
  * recent ischemic stroke (less than or equal to 14 days)
* Exclusion Criteria:

  * Less than 18 years old
  * Documented history of atrial fibrillation
  * Carotid stenosis greater than 70%
  * Pregnant women
  * Contrast allergy
  * Acute or chronic kidney disease with glomerular filtration rate<30 ml/min/1.73m2
  * Intravenous iron sensitivity
  * Serum ferritin and transferrin saturation above age-adjusted upper limit of normal. If serum ferritin is above normal, but transferrin saturation is normal, the patient is not excluded.
  * Pacemaker or other MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Vessel Wall Enhancement with Gadolinium compared to Vessel Wall Enhancement with Ferumoxytol in intracranial atherosclerosis (ICAS) group. | 1 year
  Both patient groups will have a high-resolution vessel wall enhancement-gadolinium MRI at baseline with a delayed high-resolution vessel wall enhancement-Ferumoxytol MRI. Prevalence will be analyzed between the different participants in each group.
  Hypothesis: Participants with intracranial atherosclerosis will have a high prevalence of vessel wall enhancement.

CONTACTS AND LOCATIONS:
Overall Officials: Adam de Havenon, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided